CLINICAL TRIAL: NCT05748288
Title: Development of the Virtual Unified Huntington's Disease Rating Scale
Acronym: vUHDRS
Status: Completed | Type: Observational
Sponsor: Huntington Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: vUHDRS
Record Dates: First submitted 2022-10-20; First posted 2023-02-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Personal Equipment: Participants assigned to use technology they currently own
- HSG Equipment: Participants provided technology by the sponsor

SUMMARY:
The Huntington Study Group currently holds the registered trademark for the Unified Huntington's Disease Rating Scale. The UHDRS® is a research tool which has been developed by the HSG to provide a uniform assessment of the clinical features and course of HD. The UHDRS® has undergone extensive reliability and validity testing and has been used as a major outcome measure by the HSG in controlled clinical trials.

The purpose of this research study is to determine if a standard HD assessment (the UHDRS®) is as reliable when conducted virtually as it is when conducted at an in-person visit (vUHDRS)

DETAILED DESCRIPTION:
The UHDRS® is comprised of five components:

Motor Assessment Cognitive Assessment Behavioral Assessment Independence Scale Functional Assessment Total Functional Capacity (TFC)

This observational study seeks to characterize and compare in-person versus TeleVisits. Fifty percent of participants will be provided computer equipment for their remote assessment and the other 50% will use their existing home-based equipment for this purpose.

TeleVisit is a method for participants to connect to the research study team remotely, via video and audio connection either on their computer or iPad.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female and 18 years or older at the time of signing the informed consent
2. Are able and willing to provide written informed consent
3. Are English speaking
4. Currently exhibit motor signs and symptoms of Huntington Disease
5. Have a genetic diagnosis of HD with an expanded CAG repeat (greater than or equal to 36) in the huntingtin (HTT) gene at or before Screening/Baseline visit from a validated laboratory
6. Have oral and written communication skills that are sufficient/adequate to complete all cognitive assessments
7. Are ambulatory, but may use any assistive device or require help
8. Are able to maintain stable medications for 30 days prior to Screening/Baseline through the second in-person visit
9. Have a study partner available to help with technology and set-up and to attend all study visits
10. Have the ability to get email on the device used for the study

Exclusion Criteria:

1. Are unable to complete cognitive or functional assessments due to inability to communicate
2. Are unable to obtain satisfactory internet connection (i.e., internet connection must be stable and support the audio and video needs without freezing or interruption) at home or designated location, even with provided equipment
3. Have inadequate space at home to assess 10 steps for gait assessments
4. Have active suicidal ideation endorsed with a score of 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan) if the ideation occurred within 1 year of Screening or 5 (Active Suicidal Ideation with Specific Plan and Intent) on the C-SSRS if the attempt or acts were performed within 1 year of Screening/Baseline, or participants who, in the opinion of the Site Investigator (SI), present a serious risk of suicide.
5. Have received gene therapy or an investigational drug within 30 days or 5 half-lives, whichever is longer, of the Screening/Baseline visit or plan to use an investigational drug during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from clinics with physicians who are members of the Huntington Study Group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale | from the TeleVisit to the second In-Person Visit, up to 6 weeks
  Total Motor Score:
  Minimum Score = 0 Maximum Score = 124 Higher scores indicate more impaired motor functioning
Unified Huntington's Disease Rating Scale | from the TeleVisit to the second In-Person Visit, up to 6 weeks
  Total Functional Capacity:
  Minimum Score = 0 Maximum Score = 13 Greater scores indicate higher functioning
United Huntington's Disease Rating Scale | from the TeleVisit to the second In-Person Visit, up to 6 weeks
  Independence Scale Minimum Score = 0 Maximum Score = 100 Greater scores indicate greater independence
United Huntington's Disease Rating Scale | from TeleVisit to the second In-Person Visit, up to 6 weeks
  Functional Assessment Minimum Score = 0 Maximum Score = 25 Higher scores indicate greater functionality

SECONDARY OUTCOMES:
Safety of conducting the UHDRS remotely | from initial informed consent and continue until 30 days following the Participant's completion of the study
  Reported adverse events
Unified Huntington's Disease Rating Scale | from the TeleVisit to the second In-Person Visit, up to 6 weeks
  Cognitive Function:
  Verbal Fluency minimum = 0, maximum is based upon participant responses Symbol Digit Modality (SDMT) minimum = 0, maximum = 110 Stroop minimum = 0, maximum is based upon participant responses Higher scores indicate greater cognitive function
Unified Huntington's Disease Rating Scale | Week 2, and Week 0 or Week 4
  Total Motor Score Minimum Score = 0 Maximum Score = 124 Higher scores indicate more impaired motor functioning
virtual Unified Huntington's Disease Rating Scale | from first In-Person visit through Follow-Up, up to 6 weeks
  Feasibility of completing the vUHDRS™ using participant personal equipment vs. Huntington Study Group provided equipment.
Unified Huntington's Disease Rating Scale | from the TeleVisit to the second In-Person Visit, up to 6 weeks
  Behavior minimum = 0, maximum = 88 Higher scores indicate more behavioral symptoms

OTHER OUTCOMES:
Participant Satisfaction | from first In-Person visit through Follow-Up, up to 6 weeks
  Survey

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Frank, MD, Principal Investigator — Huntington Study Group; Jody Goldstein, Study Director — Huntington Study Group
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Department of Neurology, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of South Florida, Huntington Disease Center of Excellence, Tampa, Florida
  - Northwestern University Medical Center, Department of Neurology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Hereditary Neurological Disease Center, Wichita, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Washington University, St Louis, Missouri
  - Sanford Brain and Spine Clinic, Fargo, North Dakota
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Health Science Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided